CLINICAL TRIAL: NCT03791593
Title: EVOlocumab in Stable Heart Failure With Reduced Ejection Fraction of Ischemic Etiology: EVO-HF Pilot
Acronym: EVO-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICOR-2016-05; 2017-004656-30 (EudraCT Number)
Record Dates: First submitted 2018-12-30; First posted 2019-01-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — evolocumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigators will be blinded for the biomarkers results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patient will receive evolocumab 420 mg/month on top of guideline-driven medical treatment
  Interventions: Drug: Evolocumab
- Control group (No Intervention): The patient will continue guideline-driven medical treatment

INTERVENTIONS:
Drug: Evolocumab — Evolocumab is a human IgG2 monoclonal antibody, it will add to patient treatment during 12 months.
  Other Names: Repatha
  Arms: Experimental group

SUMMARY:
Evolocumab has been able to reduce the incidence of cardiovascular events in patients that had at least one cardiovascular risk factor [28]. In patients with chronic HFrEF, as we mentioned before, treatment with statins is not recommended as it has not shown benefits in improving its prognosis. However, CAD control stands as an approach that could improve the course of the disease by preventing microlesions that further weaken the heart. A recent multicenter study, the BIOSTAT-CHF [3436], was performed to determine whether the PCSK9-LDLR axis could predict risk in patients with HF. A multivariate analysis, which included BIOSTAT risk scores, LDLR, and statin treatment as covariates, revealed a positive linear association between PCSK9 levels and the risk of mortality and the composite endpoint (death or HF-related hospitalization). A similar analysis for LDLR revealed a negative association with mortality and the composite endpoint. Future studies must assess whether PCSK9 inhibition will result in better outcomes in HF.

There is an unmet clinical need: blockade of the neurohormonal activation has provided advances in patients with HFrEF, yet mortality and morbidity remain unacceptably high. Approaching a strict control of lipid levels and CAD with evolocumab in stable HFrEF of ischemic ethology may represent a complementary pathophysiological pathway to reduce mortality and morbidity. The burden of CAD provides a solid rationale for testing the value of evolocumab in HF patients.

Therefore, a pilot trial is proposed to evaluate the beneficial effect of evolocumab by surrogate biological markers before considering an event analysis study.

Evolocumab reduces the risk of cardiovascular events in patients with established atherosclerotic disease, so this drug could play a role in HFrEF of ischemic etiology, by limiting macro- and micro-vascular coronary disease progression. In HFrEF patients due to ischemic etiology, there is a continuous troponin release due to persistent myocyte injury, which has been associated with adverse outcomes. Our hypothesis is that evolocumab may have the potential to reduce circulating hs-TnT levels, as a surrogate of myocyte injury due to atheroma progression in HFrEF. A positive result in this EVO-HF Pilot study may lead to the set-up of a large-scale multicenter prospective and randomized events study analyzing the role of lipid-lowering treatment by means of evolocumab in HFrEF of ischemic etiology

DETAILED DESCRIPTION:
Evolocumab has been able to reduce the incidence of cardiovascular events in patients that had at least one cardiovascular risk factor [28]. In patients with chronic HFrEF, as we mentioned before, treatment with statins is not recommended as it has not shown benefits in improving its prognosis. However, CAD control stands as an approach that could improve the course of the disease by preventing microlesions that further weaken the heart. A recent multicenter study, the BIOSTAT-CHF [3436], was performed to determine whether the PCSK9-LDLR axis could predict risk in patients with HF. A multivariate analysis, which included BIOSTAT risk scores, LDLR, and statin treatment as covariates, revealed a positive linear association between PCSK9 levels and the risk of mortality and the composite endpoint (death or HF-related hospitalization). A similar analysis for LDLR revealed a negative association with mortality and the composite endpoint. Future studies must assess whether PCSK9 inhibition will result in better outcomes in HF.

There is an unmet clinical need: blockade of the neurohormonal activation has provided advances in patients with HFrEF, yet mortality and morbidity remain unacceptably high. Approaching a strict control of lipid levels and CAD with evolocumab in stable HFrEF of ischemic ethology may represent a complementary pathophysiological pathway to reduce mortality and morbidity. The burden of CAD provides a solid rationale for testing the value of evolocumab in HF patients.

Evolocumab reduces the risk of cardiovascular events in patients with established atherosclerotic disease, so this drug could play a role in HFrEF of ischemic etiology, by limiting macro- and micro-vascular coronary disease progression. In HFrEF patients due to ischemic etiology, there is a continuous troponin release due to persistent myocyte injury, which has been associated with adverse outcomes. Our hypothesis is that evolocumab may have the potential to reduce circulating hs-TnT levels, as a surrogate of myocyte injury due to atheroma progression in HFrEF. A positive result in this EVO-HF Pilot study may lead to the set-up of a large-scale multicenter prospective and randomized events study analyzing the role of lipid-lowering treatment by means of evolocumab in HFrEF of ischemic etiology.

Therefore, a pilot trial is proposed to evaluate the beneficial effect of evolocumab by surrogate biological markers before considering an event analysis study.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent
2. Patient ≥18 years and ≤80 years of age
3. LVEF <40%
4. Ischemic etiology (evidence of at least one acute coronary event and/or CAD by coronary angiography or multi slice CT)
5. New York Heart Association (NYHA) class II
6. NT-proBNP ≥ 400 pg/mL
7. Hs-TnT >10 pg/mL
8. LDL ≥ 70 mg/dL
9. Stable CAD (last ACS before the last 3 months)
10. GDMT according to 2016 ESC HF guidelines for at least the last 3 months.
11. Statin treatment, whichever dose the patient receives at the time of enrolment, stable for at least 1 month, without need to statin uptitration.

Exclusion Criteria:

1. Extracardiac disease with estimated life expectancy less than 1 year
2. Contraindication to receiving evolocumab
3. Hypersensitivity to the active substance or to any of the excipients
4. Female subject who has not used an acceptable method of birth control for at least 1 month prior to screening and/or is not willing to inform her partner of her participation in this clinical trial and to use an acceptable method of effective birth control during treatment with evolocumab and for an additional 15 weeks after the end of treatment with evolocumab, unless the female subject is permanently sterilized or postmenopausal:

   A female is considered of childbearing potential unless permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or postmenopausal with menopause defined as:
   * Age ≥55 years and ≥12 months of spontaneous and continuous amenorrhea, or
   * Age <55 years but no spontaneous menses for ≥2 years, or
   * Age <55 years and spontaneous menses within the past 1 year, but currently amenorrheic, AND with follicle-stimulating hormone (FSH) levels >40 IU/L or estradiol levels <5 ng/dL or according to the definition of "postmenopausal range" for the laboratory involved.
5. Patient <18 or ≥ 81 years
6. Liver dysfunction (AST or ALT> 3 times the upper limit of normal value).
7. Severe renal dysfunction (estimated glomerular filtration rate [eGFR] < 30 ml/min/1.73m²) or renal replacement therapy at screening (CKD-EPI equation).
8. Coronary revascularization in the 3 months prior to randomization or pending coronary revascularization.
9. Previous haemorrhagic stroke
10. Uncontrolled hypertension (systolic blood pressure ≥ 140 or/and diastolic blood pressure ≥ 90 mmHg) either on or off therapy at screening or at baseline
11. Uncontrolled hypothyroidism or hyperthyroidism
12. Type 1 diabetes; newly diagnosed or poorly controlled type 2 diabetes (HbA1c > 8.5%)
13. Uncontrolled cardiac arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in hs-TnT levels at 1 year | at 12 months of follow-up
  Change of high-sensitivity troponin T (hs-TnT) levels from baseline to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Bayes-Genís, MD,PhD,FESC, Principal Investigator — HUGTIP
Locations (3):
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia